CLINICAL TRIAL: NCT04646668
Title: Comparative Abuse Liability of Cigarettes, E-cigarettes, and Heat-not-burn Devices Among African American and White Smokers
Brief Title: Comparative Abuse Liability Among African American and White Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 00145421
Record Dates: First submitted 2020-11-09; First posted 2020-11-30 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: 1. 20 eligible African American and white smokers will be randomized. A 1:1 randomization to product order (combustible cigarette, e-cigarette, heat-not-burn vs. combustible cigarette, heat-not-burn, e-cigarette). Randomization will be determined by computer-generated random numbers. Randomization assignments will be placed in sealed envelopes with sequential study identification numbers. After baseline data collection has been completed, the research assistant will select the sequential study identification number to determine the randomization assignment
  2. No blinding is involved.
  3. Due to the pilot nature of the current study, formal power calculations were not conducted. ANOVAs will be conducted to detect within-subject differences between products. A Bonferroni correction will be applied to adjust for multiple comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- E-Cigarette then Heat not burn. (Active Comparator): We will use a 1:1 fashion randomization to product order (combustible cigarette, e-cigarette, heat-not-burn device.
  Interventions: Combination Product: E-cigarette and Heat not burn
- Heat not burn then E-Cigarette (Active Comparator): We will use a 1:1 fashion randomization to product order combustible cigarette, heat-not-burn device, e-cigarette.
  Interventions: Combination Product: E-cigarette and Heat not burn

INTERVENTIONS:
Combination Product: E-cigarette and Heat not burn — Current smokers will be randomized to session order and complete a standardized 10-puff bout (5 minutes) followed by a 60-minute ad libitum session with each product (usual brand cigarette, e-cigarette, heat-not-burn).

SUMMARY:
The study is a randomized crossover trial. Current smokers will complete a session with each product: usual brand cigarette, e-cigarette, and heat-not-burn. The objective of this survey is to assess for ongoing use of study products and is part of safety monitoring.

DETAILED DESCRIPTION:
The study is a randomized crossover trial. Current smokers will be randomized to session order and complete a standardized 10-puff bout (5 minutes) followed by a 60-minute ad libitum session with each product (usual brand cigarette, e-cigarette, heat-not-burn). Throughout each visit, blood will be collected for nicotine analysis via an IV catheter placed in the patient's arm. Blood samples will be aliquoted into two separate vials. One will be analyzed for the current study and one will be placed in a biospecimen repository if participant provides consent for biorepository. Puff topography will be collected passively throughout the session to measure puffing patterns. Participants will complete self-report measures of nicotine withdrawal and craving. Finally, breath samples will be collected to measure changes in exhaled carbon monoxide, a potent lung toxicant, pre- and post-product use. At the final visit, participants will complete a behavioral economics concurrent choice task (see below for description) to behaviorally measure their decisions regarding use of e-cigarettes or heat not burn products in place of cigarettes. Finally, participants will be contacted by phone 6 months following the conclusion of visit 3 (or study discontinuation) to complete a phone survey. The objective of this survey is to assess for ongoing use of study products and is part of safety monitoring. We have no hypotheses related to the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic African American or white/Caucasian,
* ≥21 years old, smoke 5-30 cigarettes per day,
* daily cigarette smoker
* smoked at current rate for at least 6 months
* interested in trying e-cigarettes and heat not burn products
* not interested in or unable/unwilling to quit cigarette smoking
* willing to complete three in-person study visits
* willing to have IV catheter placed

Exclusion Criteria:

* Interested in quitting cigarettes in the next 30 days
* use of smoking cessation pharmacotherapy in the past 30 days
* use of non-cigarette tobacco products in the past 30 days
* use of e-cigarettes >5x in lifetime
* use of e-cigarettes ≥4 of the past 30 days
* use of heat not burn products >5x in lifetime
* use of heat not burn products ≥4 of the past 30 days
* weight < 110 lbs
* uncontrolled hypertension (systolic BP ≥ 180 or diastolic BP ≥ 105)
* pregnant, plans to become pregnant, or breastfeeding
* live >10 miles from study site (Fairway CRU)
* current enrollment is a research study or program that aims to alter tobacco use

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Leavens, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Funk OL, Nollen NL, Wagener TL, Ahluwalia JS, Mayo MS, Mahmud KMF, Lambart L, Leavens ELS. Concurrent Choice Assessment of Preference and Substitutability of E-cigarettes and Heated Tobacco Products for Combustible Cigarettes Among African American and White Smokers. Nicotine Tob Res. 2023 Jul 14;25(8):1505-1508. doi: 10.1093/ntr/ntad052. PMID 37042345

RESULTS

PARTICIPANT FLOW:
Groups:
- Cigarette, E-Cigarette Then Heat Not Burn.: At lab visit 1 participants receive their usual brand cigarette during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Following at least a 48-hour washout period, at lab visit 2, participants receive electronic cigarette during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Following at least a 48-hour washout period, at lab visit 3, participants receive Heat Not Burn during the 10-puff standardized puff bout and 60-minute ad libitum session.
- Cigarette, Heat Not Burn Then E-Cigarette: At lab visit 1 participants receive their usual brand cigarette during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Following at least a 48-hour washout period, at lab visit 2, participants receive Heat Not Burn during the 10-puff standardized puff bout and 60-minute ad libitum session.
  Following at least a 48-hour washout period, at lab visit 3, participants receive electronic cigarette during the 10-puff standardized puff bout and 60-minute ad libitum session.
Period: Overall Study
Arm/Group | Cigarette, E-Cigarette Then Heat Not Burn. | Cigarette, Heat Not Burn Then E-Cigarette
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline blood plasma nicotine concentration
Groups:
- Total: Total of all reporting groups
Arm/Group | Cigarette, E-Cigarette Then Heat Not Burn. | Cigarette, Heat Not Burn Then E-Cigarette | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [24 to 65] | 54.1 [34 to 65] | 54.1 [24 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Delivery
Description: Blood plasma nicotine concentration after 10 puff bout of product at 5 minutes
Time Frame: Baseline, after 10 puff bout of product at 5 minutes
Population: Blood plasma nicotine concentration 5 minutes after start
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Cigarette: Participants used their own brand cigarette during the first study visit.
- E-Cigarette: Participants who used the e-cigarette product during either the second or third study visit.
- Heat Not Burn: Participants who used the heat not burn product during either the second or third study visit.
Arm/Group | Cigarette | E-Cigarette | Heat Not Burn
Number analyzed (Participants) | 21 | 21 | 21
ng/mL | 14.13 [4.3 to 35.6] | 6.79 [0.5 to 26.6] | 9.15 [1.5 to 22.5]
Statistical Analysis 1: Comparison: Cigarette vs E-Cigarette vs Heat Not Burn; The null hypothesis is that there is no difference in nicotine delivery between cigarettes, e-cigarettes, and heat not burn after the standardized 10-puff bout. ANOVAs were conducted to detect differences between products for nicotine concentration at five minutes (immediately following 10-puff bout). The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority — Due to the pilot nature of the current study, formal power calculations were not conducted; p = 0.002, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Description: No differences in definitions.
Groups:
- Cigarette: At the first visit, all participants used their usual brand of cigarette.
  Participants completed a standardized 10-puff bout (5 minutes) followed by a 60-minute ad libitum session with cigarettes.
- E-Cigarette: At the second and third visits, participants were randomly assigned either e-cigarette or heat not burn. All participants completed a visit for each product but the order was random.
  Participants completed a standardized 10-puff bout (5 minutes) followed by a 60-minute ad libitum session with the e-cigarette.
- Heat Not Burn: At the second and third visits, participants were randomly assigned either e-cigarette or heat not burn. All participants completed a visit for each product but the order was random.
  Participants completed a standardized 10-puff bout (5 minutes) followed by a 60-minute ad libitum session with heat-not-burn.
Arm/Group | Cigarette | E-Cigarette | Heat Not Burn
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04646668/Prot_SAP_000.pdf